CLINICAL TRIAL: NCT06000995
Title: Determination of Fiberoptic Bronchoscopy Sedation Protocols; Survey Study on Sedation Attitudes and Behaviors of Chest Diseases Specialists in Turkey
Brief Title: Determination of Fiberoptic Bronchoscopy Sedation Protocols in Turkey
Status: Completed | Type: Observational
Sponsor: Samsun University (Other)
Responsible Party: Principal Investigator, dilan akyurt, Principle investigator, Samsun University
Other Study IDs: B.30.2.ODM.0.20.08/340
Record Dates: First submitted 2023-07-29; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Fiberoptic Bronchoscopy
Keywords: sedation; non-operating room anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Pulmonologists: pulmonologists actively performing fiberoptic bronchoscopy
  Interventions: Other: Survey Questions

INTERVENTIONS:
Other: Survey Questions — Thirty questions generally consist of three parts; In the first part, there are 8 questions containing the personal information of the doctors (age, gender, title, institution, etc.). In the second part, 13 questions were included in order to make a general assessment such as the sedative agents used by the doctors before and during the bronchoscopy procedure and the satisfaction with the sedative method used. In the third part, 9 questions were given to determine the preferred follow-up methods during the procedure.

SUMMARY:
Fiberoptic bronchoscopy (FOB), which is difficult to tolerate while awake, is recommended to be performed by the patient under sedation. The aim of this study is to determine the attitudes and behaviors of chest diseases specialists who do FOB in Turkey about sedation with a 30-question online questionnaire.

DETAILED DESCRIPTION:
Fiberoptic bronchoscopy is the imaging of the tracheobronchial tree for diagnosis and treatment in lung diseases. The operation performed through the airway is difficult for the patient to tolerate. Therefore, it is recommended to perform the procedure under sedation. With this survey study, it was aimed to determine the sedation protocols preferred by pulmonologists who perform active fiberoptic bronchoscopy throughout Turkey during the procedure.

Thirty questions were determined for the questionnaire to be used as a data collection method by the researchers. The questions generally consist of three parts; In the first part, there are 8 questions containing the personal information of the doctors (age, gender, title, institution, etc.). In the second part, 13 questions were included in order to make a general assessment such as the sedative agents used by the doctors before and during the bronchoscopy procedure, and the satisfaction with the sedative method used. In the third part, 9 questions were given to determine the preferred follow-up methods during the procedure. The questions are designed to be presented to participants over the network using google forms.

ELIGIBILITY:
Inclusion Criteria:

* Currently working as a pulmonologist

Exclusion Criteria:

* Not actively performing fiberoptic bronchoscopy for the past five years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pulmonologists who are still working in Turkey and have been actively doing FOB for the last 5 years
Sampling Method: Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
FOB related survey questions | 15 minutes
  The pulmonologists' responses to 30 questionnaire questions were recorded. Thirty questions generally consisted of three parts; Part 1; personal information of doctors (age, gender, title, institution, etc.), in section 2; sedative agents used by doctors before and during bronchoscopy and satisfaction with the sedative method used, part 3; preferred follow-up methods during the procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Dilan Akyurt, Samsun, Turkey (Türkiye)

REFERENCES:
- [Background] Wahidi MM, Jain P, Jantz M, Lee P, Mackensen GB, Barbour SY, Lamb C, Silvestri GA. American College of Chest Physicians consensus statement on the use of topical anesthesia, analgesia, and sedation during flexible bronchoscopy in adult patients. Chest. 2011 Nov;140(5):1342-1350. doi: 10.1378/chest.10-3361. PMID 22045879
- [Background] Du Rand IA, Blaikley J, Booton R, Chaudhuri N, Gupta V, Khalid S, Mandal S, Martin J, Mills J, Navani N, Rahman NM, Wrightson JM, Munavvar M; British Thoracic Society Bronchoscopy Guideline Group. British Thoracic Society guideline for diagnostic flexible bronchoscopy in adults: accredited by NICE. Thorax. 2013 Aug;68 Suppl 1:i1-i44. doi: 10.1136/thoraxjnl-2013-203618. No abstract available. PMID 23860341
- [Background] Gaisl T, Bratton DJ, Heuss LT, Kohler M, Schlatzer C, Zalunardo MP, Frey M, Franzen D. Sedation during bronchoscopy: data from a nationwide sedation and monitoring survey. BMC Pulm Med. 2016 Aug 5;16(1):113. doi: 10.1186/s12890-016-0275-4. PMID 27495824
- [Background] Hautmann H, Hetzel J, Eberhardt R, Stanzel F, Wagner M, Schneider A, Dirschinger R, Poszler A. Cross-Sectional Survey on Bronchoscopy in Germany--The Current Status of Clinical Practice. Pneumologie. 2016 Feb;70(2):110-6. doi: 10.1055/s-0041-110288. Epub 2016 Feb 19. PMID 26894392